CLINICAL TRIAL: NCT03288740
Title: A Single-centre, Randomised, Double-blind, Placebo-controlled, Multiple-dose Trial to Assess the Pharmacokinetics, Safety and Tolerability of Semaglutide in Healthy Chinese Subjects
Brief Title: A Trial to Assess the Pharmacokinetics, Safety and Tolerability of Semaglutide in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9535-3686; U1111-1149-6572 (Other: World Health Organization (WHO))
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Semaglutide 0.5 mg (Experimental): Participants will enter a 13 weeks treatment with 4 weeks dosing at dose level 0.25 mg and 9 weeks at 0.5 mg semaglutide.
  Interventions: Drug: Semaglutide 0.5 mg
- Semaglutide 0.5 mg placebo (Placebo Comparator): Participants will enter a 13 weeks treatment with 4 weeks dosing at dose level 0.25 mg and 9 weeks at 0.5 mg semaglutide placebo.
  Interventions: Drug: Placebo (semaglutide 0.5 mg)
- Semaglutide 1.0 mg (Experimental): Participants will have 13 weeks treatment with 4 weeks dosing at dose level of 0.25 mg, 4 weeks at 0.5 mg, and 5 weeks at 1.0 mg semaglutide.
  Interventions: Drug: Semaglutide 1.0 mg
- Semaglutide 1.0 mg placebo (Placebo Comparator): Participants will have 13 weeks treatment with 4 weeks dosing at dose level of 0.25 mg, 4 weeks at 0.5 mg, and 5 weeks at 1.0 mg semaglutide placebo.
  Interventions: Drug: Placebo (semaglutide 1.0 mg)

INTERVENTIONS:
Drug: Semaglutide 0.5 mg — A dose of 0.25 mg semaglutide gradually increased to 0.5 mg injected subcutaneously (under the skin) once weekly for 13 weeks.
  Arms: Semaglutide 0.5 mg
Drug: Placebo (semaglutide 0.5 mg) — A dose of 0.25 mg semaglutide placebo gradually increased to 0.5 mg injected subcutaneously (under the skin) once weekly for 13 weeks.
  Arms: Semaglutide 0.5 mg placebo
Drug: Semaglutide 1.0 mg — A dose of 0.25 mg semaglutide gradually increased to 1.0 mg injected subcutaneously (under the skin) once weekly for 13 weeks.
  Arms: Semaglutide 1.0 mg
Drug: Placebo (semaglutide 1.0 mg) — A dose of 0.25 mg semaglutide placebo gradually increased to 1.0 mg injected subcutaneously (under the skin) once weekly for 13 weeks.
  Arms: Semaglutide 1.0 mg placebo

SUMMARY:
The main purpose of the trial is to assess the pharmacokinetics of semaglutide (i.e. the way the drug is distributed in the body over a period of time) following once-weekly administration of semaglutide in healthy Chinese subjects. Different dose levels (0.5 and 1.0 mg) will be investigated in this trial. Participants will be administered semaglutide or placebo once-weekly by subcutaneous injection (under the skin fold of the abdominal wall) using a pen injector with a very small, thin needle by the trial doctor at the trial site for 13 weeks. The trial consists of 23 visits in total, including visit for screening and safety tests, visit for dose administration and blood sample collection. The total time of participation will be approximately 18-22 weeks depending on participant's individual visit schedule.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female Chinese subjects
* Age between 18 to 55 years (both inclusive) at the time of signing informed consent
* Body mass index (BMI) between 20 and 24.9 kg/sqm (both inclusive)
* Body weight greater than or equal to 54.0 kg

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential not using an adequate contraceptive method throughout the trial including follow-up period. Adequate contraceptive measures are sterilisation, intrauterine device (IUD), oral contraceptives or barrier methods
* Any clinically significant disease history, in the opinion of the investigator, or systemic or organ disease including: pulmonary, gastrointestinal, hepatic, neurologic, renal, genitourinary and endocrine, dermatologic or hematologic diseases
* Use of prescription or non-prescription systemic products (including routine or non-routine vitamins or herbal products) or topical medicinal products (except paracetamol and oral contraceptives) within 3 weeks (or within 5 half-lives of the medicinal product, whichever is longest) prior to Visit 2 (randomisation)
* Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2
* History of pancreatitis (acute or chronic)
* Calcitonin greater than or equal to 50 ng/L
* Blood donation, surgery or trauma with significant blood loss (400 mL) within the last 12 weeks prior to screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-08-07 (Actual)

PRIMARY OUTCOMES:
Area under the semaglutide plasma concentration time curve at steady state (semaglutide 0.5 mg) | 0-168 hours after last administration of semaglutide
  Calculated based on semaglutide measured in blood.
Area under the semaglutide plasma concentration time curve at steady state (semaglutide 1.0 mg) | 0-168 hours after last administration of semaglutide
  Calculated based on semaglutide measured in blood.

SECONDARY OUTCOMES:
Maximum observed semaglutide plasma concentration at steady state | 0-168 hours after last administration of semaglutide
  Calculated based on semaglutide measured in blood.
Time to maximum observed semaglutide plasma concentration at steady state | 0-168 hours after last administration of semaglutide
  Calculated based on semaglutide measured in blood.
Total apparent clearance of semaglutide at steady state | 0-168 hours after last administration of semaglutide
  Calculated based on semaglutide measured in blood.
Terminal elimination half-life of semaglutide at steady state | 0-840 hours after last administration of semaglutide
  Calculated based on semaglutide measured in blood.
Apparent volume of distribution of semaglutide at steady state | 0-840 hours after last administration of semaglutide
  Calculated based on semaglutide measured in blood.
Trough plasma semaglutide concentration | Before dosing at day 29, 57, 78, 85 and 92
  Calculated based on semaglutide measured in blood.
Dose-corrected accumulation ratio | Based on the area under the semaglutide plasma concentration curve from 0-168 hours after the first dose and the area under the semaglutide plasma concentration curve 0-168 hours after the last dose
  Calculated based on semaglutide measured in blood.
Area under the semaglutide plasma concentration time curve | 0-168 hours after the first dose of semaglutide 0.25 mg (starting dose level)
  Calculated based on semaglutide measured in blood.
Maximum observed semaglutide plasma concentration | 0-168 hours after the first dose of semaglutide 0.25 mg (starting dose level)
  Calculated based on semaglutide measured in blood.
Time to maximum observed semaglutide plasma concentration | 0-168 hours after the first dose of semaglutide 0.25 mg (starting dose level)
  Calculated based on semaglutide measured in blood.
Number of treatment emergent adverse events (TEAEs) | Visit 2 (Day 1) - visit 23 (Day 120-127)
  Count and % of adverse events
Number of hypoglycaemic episodes | Visit 2 (Day 1) - visit 23 (Day 120-127)
  Count of episodes
Incidence of anti-semaglutide antibodies (positive/negative) at follow-up | Visit 23 (Day 120-127)
  Count of episodes

CONTACTS AND LOCATIONS:
Locations (1):
- Novo Nordisk Investigational Site, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Result] Shi A, Xie P, Nielsen LL, Skjoth TV, He X, Haugaard SP. Pharmacokinetics, Safety and Tolerability of Once-Weekly Subcutaneous Semaglutide in Healthy Chinese Subjects: A Double-Blind, Phase 1, Randomized Controlled Trial. Adv Ther. 2021 Jan;38(1):550-561. doi: 10.1007/s12325-020-01548-y. Epub 2020 Nov 7. PMID 33159658